CLINICAL TRIAL: NCT05043597
Title: Effectiveness Evaluation in Thrombus Aspiration in Patients With STEMI and High Thrombotic Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LHD Thrombus aspiration
Record Dates: First submitted 2021-08-25; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrombus aspiration (Experimental)
  Interventions: Procedure: Thrombus aspiration
- control group (No Intervention)

INTERVENTIONS:
Procedure: Thrombus aspiration — Thrombus aspiration
  Arms: Thrombus aspiration

SUMMARY:
This study intends to evaluate thrombus on the basis of different methods for evaluating thrombus load The effect of aspiration on the prognosis of STEMI patients with high thrombotic load Provide a basis for the standardized use of aspiration; at the same time, discover the best benefit groups for thrombus aspiration

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years; (2) Voluntary signing of informed consent; (3) Onset of 12 hours STEMI patients who underwent PCI reperfusion therapy within time; (4) The guidewire passes through the lesion and the blood Heavy embolism load (TIMI thrombus classification ≥ 3).

Exclusion Criteria:

* (1) Hemodynamics is unstable or there is cardiogenic shock; (2) After thrombolytic therapy; (3) The expected survival time is less than 6 months due to non-cardiac diseases; (4) Past trips Coronary artery bypass graft patients; (5) Participate in other drug and device research within 30 days; (6) Before surgery, clear active gastrointestinal bleeding or other contraindications for taking dual antiplatelet drugs (7) Patients deemed unsuitable for enrollment by other researchers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3838 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse cardiovascular events | 3 years
  Including cardiogenic death, recurring myocardial infarction Stent thrombosis or target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, China